CLINICAL TRIAL: NCT03005418
Title: A Phase 2/3 Study for the Evaluation of Safety and Efficacy of Humacyte's Human Acellular Vessel for Vascular Replacement or Reconstruction in Patients With Life or Limb-threatening Vascular Trauma
Brief Title: Humacyte Human Acellular Vessel (HAV) in Patients With Vascular Trauma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: Atlantic Research Group (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V005
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Trauma; Vascular System Injury
MeSH Terms: conditions — Wounds and Injuries; Vascular System Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Human Acellular Vessel (HAV) (Experimental): Patients with life or limb threatening traumatic injury to an arterial vessel in the limb or torso, other than the heart, will be implanted with the Humacyte Human Acellular Vessel (HAV) as an interposition vessel or bypass using standard vascular surgical techniques.
  Interventions: Biological: Human Acellular Vessel (HAV)

INTERVENTIONS:
Biological: Human Acellular Vessel (HAV) — The investigational medicinal product (IMP) - the Human Acellular Vessel (HAV) is a sterile acellular tubular graft composed of human collagen types I and III and other extracellular matrix proteins, including fibronectin and vitronectin which can be used for arterial bypass or reconstruction in patients with life or limb threatening vascular trauma. The vessel is 6 mm in diameter and approximately 42 cm in length. The product is supplied on a silicone mandrel immersed in sterile phosphate buffered saline in a sealed and labeled plastic container. The Humacyte HAV is implanted using standard vascular surgical techniques similar to placement of predicate peripheral vascular prostheses.

SUMMARY:
This study evaluates the use of the Human Acellular Vessel (HAV) in adults with vascular trauma below the neck who are undergoing vascular reconstructive surgery. There will be a torso cohort and a limb cohort. All subjects will be implanted with a HAV as an interposition vessel or bypass using standard vascular surgical techniques. There is no control arm.

DETAILED DESCRIPTION:
This is a prospective, multicenter, multi cohort, non-randomized phase 2 study in up to 40 adult patients with life or limb threatening vascular trauma which requires surgical repair. There will be a limb cohort and a torso cohort. The limb cohort will include patients who require repair of a vessel contained to the upper or lower extremity. The torso cohort includes patients who require repair of vessels within the thorax (excluding the heart), abdomen, and retroperitoneum. Subjects will be implanted with a Humacyte Human Acellular Vessel (HAV) as an interposition vessel or bypass using standard vascular surgical techniques. There is no control arm.

The active study duration for each study participant will be 36 months from HAV implantation or until HAV failure/ removal/ death if earlier. Follow up after month 12 will involve the capture of information on assessments performed at "standard of care" routine clinic visits or by telephone follow up with the patient or his/her physician with physical exam and ultrasound at month 24 and month 36

The total expected duration of the clinical study is 61 months (24 months of enrollment and 36 months of follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with life or limb threatening traumatic injury to an arterial vessel in the limb or torso, other than the heart, which requires replacement or reconstruction
2. Preoperative imaging or clinical examination indicates the damaged vessel has a defect length of ≤ 38cm and is appropriately size matched to the 6mm Human Acellular Vessel (HAV) per the judgment of the treating surgeon taking into account vasoconstriction and situational inflow and outflow considerations.
3. Autologous vein graft is either not feasible in the judgment of the treating surgeon (e.g. because of lack of availability of suitable conduit, presence of severe venous insufficiency) or is not desirable because of the urgency of revascularization
4. Aged 18 to 85 years old, inclusive
5. Able to communicate meaningfully with investigative staff, and able to comply with entire study procedures. If the patient is unconscious, then information from a reliable witness indicates that the patient would normally be able to comply with study procedures
6. Patient or relative is able, willing and competent to give informed consent
7. Life expectancy of at least 1 year

Exclusion Criteria:

1. Mangled Extremity Severity Score (MESS) of ≥ 7
2. Limb at high risk of amputation despite vascular reconstruction (e.g., because of crush injury)
3. Catastrophic injuries that make survival unlikely (e.g. Abbreviated Injury Scale (AIS) > 5 or Injury Severity Score (ISS) >60)
4. HAV may not be used for coronary artery repair
5. Known pregnant women
6. Known medical condition which would preclude long term antiplatelet therapy after resolution of acute injuries
7. Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the HAV
8. Previous exposure to HAV
9. Known participation in any investigational study within the last 30 days
10. Employees of the sponsor or patients who are employees or relatives of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
HAV primary patency | 30 days
  Primary patency is defined as 'the interval from the time of access placement until any intervention designed to maintain or reestablish patency, access thrombosis or the measurement of patency', i.e., patent without interventions
Frequency and Severity of Adverse Events | 36 months

SECONDARY OUTCOMES:
Limb viability (avoidance of amputation; limb cohort only) | 36 months
HAV primary patency | 36 months
  Primary patency is defined as 'the interval from the time of access placement until any intervention designed to maintain or reestablish patency, access thrombosis or the measurement of patency', i.e., patent without interventions
HAV primary assisted patency | 36 months
  Primary assisted patency is defined as 'the interval from the time of access placement until access thrombosis or the time of measurement of patency, including intervening manipulations (surgical or endovascular interventions) designed to maintain the functionality of patent access' i.e., patent without an intervention to clear a thrombus
HAV secondary patency | 36 months
  Secondary patency is defined as 'the interval from the time of access placement until access abandonment', i.e., patent with or without interventions
Rate of HAV interventions | 36 months
Patient survival | 36 months
HAV remodeling as shown by histopathology of any clinical explants | 36 months
Frequency of anastomotic bleeding or spontaneous rupture | 36 months
Frequency of HAV infection | 36 months
Frequency of HAV thrombosis | 36 months
Frequency of HAV pseudoaneursym formation | 36 months
Frequency of HAV aneursym formation | 36 months
Frequency of HAV of hemodynamically significant stenosis (>70% by duplex ultrasound criteria) | 36 months
Frequency of HAV removal | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, MD, Study Director — Humacyte, Inc.
Locations (32):
- United States (28):
  - Jacob Medical Center at UC San Diego, La Jolla, California
  - Keck Hospital of University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Cener, Los Angeles, California
  - UCI Medical Center, Orange, California
  - University California, Davis, Sacramento, California
  - University of California San Diego (UCSD) Medical Center, San Diego, California
  - Ernest E Moore Shock Trauma Center at Denver Health, Denver, Colorado
  - UF Health Jacksonville, Jacksonville, Florida
  - Jackson South Medical Center, Miami, Florida
  - Ryder Trauma Center, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - R Adams Cowley Baltimore Shock Trauma, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University (SLU), St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Duke University Hospital, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas - Dell Medical School, Austin, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Israel (4):
  - Soroka Medical Center - Vascular Surgery Department, Beersheba
  - Rambam Health Care Campus - Vascular Surgery Department, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - The Chaim Sheba Medical Center - Vascular Surgery Department, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lum Y, Moore EE, Kundi R, Morrison J, Shores JT, Niklason LE, Parikh S. Bioengineered human blood vessels to treat hospital-acquired vascular complications. J Vasc Surg Cases Innov Tech. 2025 Sep 8;11(6):101976. doi: 10.1016/j.jvscit.2025.101976. eCollection 2025 Dec. PMID 41140335
- [Derived] Moore EE, Curi M, Namias N, Kundi R, Lum YW, Fox CJ, Rajani RR, Rasmussen TE, Sokolov O, Niklason LE, Khondker Z, Parikh SJ; CLN-PRO-V005 Investigators and the CLN-PRO-V017 Investigators. Bioengineered Human Arteries for the Repair of Vascular Injuries. JAMA Surg. 2025 Feb 1;160(2):181-189. doi: 10.1001/jamasurg.2024.4893. PMID 39565635